CLINICAL TRIAL: NCT03879512
Title: Autologous Dendritic Cells and Metronomic Cyclophosphamide in Combination With Checkpoint Blockade for Relapsed High-Grade Gliomas in Children and Adolescents
Brief Title: Autologous Dendritic Cells, Metronomic Cyclophosphamide and Checkpoint Blockade in Children With Relapsed HGG
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIT-HGG Rez Immunovac
Record Dates: First submitted 2019-03-12; First posted 2019-03-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-12

CONDITIONS: Childhood Glioblastoma
Keywords: cancer vaccine; high-grade glioma; immunomodulation; checkpoint blockade
MeSH Terms: conditions — Astrocytoma; Glioma | interventions — Reoperation; Cancer Vaccines; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active vaccination arm (Experimental): All patients receive depletion of regulatory T cells, reoperation, followed by a personalized cancer vaccine and double checkpoint blockade.
  Interventions: Drug: depletion of regulatory T cells; Procedure: reoperation; Biological: cancer vaccine; Biological: checkpoint blockade

INTERVENTIONS:
Drug: depletion of regulatory T cells — oral metronomic cyclophosphamide
Procedure: reoperation — resection of relapsed tumor in order to improve clinical condition of the patient and to acquire tumor tissue for vaccine generation
Biological: cancer vaccine — 4 weekly intradermal injections of lysate-loaded dendritic cells, followed by 3 monthly boost vaccines with tumor lysate and further boost vaccines every three months
Biological: checkpoint blockade — Immediately one week after the DC-induction vaccines, patients will receive four applications of Nivolumab/Ipilimumab double checkpoint blockade in threeweekly intervals, followed by Nivolumab monotherapy every month for a total duration of one year.

SUMMARY:
This phase I/II trials evaluates the feasibility, safety and efficacy of an individualized cancer vaccine, based on autologous, tumor-lysate loaded dendritic cells in children and adolescents with relapsed high-grade gliomas. In addition, regulatory T cells are depleted by a short cycle of metronomic cyclophosphamide upfront of the vaccine in order to facilitate induction of immune responses.

Therapeutic DC vaccines are followed by four cycles of Nivo/Ipi double checkpoint blockade and a Nivolumab monotherapy maintenance in order to optimize the induced T-cell response.

DETAILED DESCRIPTION:
Relapsed high-grade gliomas (in the following addressed as high-grade gliomas = HGG) in children and adolescents represent a very bad prognosis group for which a recommended standard salvage therapy is currently not available.

Combination of Dendritic Cell (DC) vaccination, metronomic cyclophosphamide, and checkpoint blockade will be investigated in the present trial as a new treatment strategy for these patients: metronomic cyclophosphamide has been shown to significantly reduce numbers of regulatory T cells (Treg) without inducing general leukopenia. DCs might induce tumour-directed immune responses thereby facilitating long-term remissions. Efficacy of primed T-cell responses by the vaccine will potentially be enhanced by the application of checkpoint inhibitors Nivolumab (antiPD-L1) and Ipilimumab (antiCTLA4) in the post-vaccine phase and during maintenance.

Cyclophosphamide is an established drug used as an anti-cancer or immunosuppressive substance since decades, with extensive experience when used in low, non-myeloablative dosages. DCs represent an innovative new strategy in cellular immunotherapy. DCs in cancer patients have been used in a number of smaller studies, and in some of these trials, promising results could be obtained. Several studies showed a trend towards a prolonged overall survival with a few long-term survivors which is otherwise extremely rare in this high-risk population. Results seemed to be more favourable in pediatric than in adult patients. Checkpoint inhibitors (antiPD-L1 and/or antiCTLA4) have been shown to exhibit synergistic effects with vaccines in preclinical models, and prelimnary data of several early stage trials have shown promising results. Therefore, our study aims to improve the efficacy of a DC-based therapeutic vaccine by optimizing the conditions upfront of the vaccine (Treg depletion) and improving T-cell responses by checkpoint blockade after the vaccine in the effector phase.

In conclusion, this study will exploit the optimal efficacy of a therapeutic vaccine in children and adolescents with relapsed HGG.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of relapsed high-grade malignant glioma confirmed by central neuropathological and neuroradiological review (last magnetic resonance imaging diagnosis not older than 4 weeks) - including glioblastoma multiforme (WHO IV), anaplastic astrocytoma World Health Organization (WHO III), anaplastic oligodendroglioma (WHO III), anaplastic oligoastrocytoma (WHO III), anaplastic pilocytic astrocytoma (WHO III), anaplastic ganglioglioma (WHO III), anaplastic pleomorphic xanthoastrocytoma (analogous to WHO III), giant cell glioblastoma (WHO IV), and gliosarcoma (WHO IV) relapsed after first-line therapy.
2. Patients aged 3 years and older but under 21 years at time of relapse diagnosis
3. Written informed consent of the patient (mandatory from 14 years of age) or the parents (mandatory till 18 years of age).
4. Prospect of resection of relapse tumour by neurosurgery (total, subtotal or partial)

Exclusion Criteria:

1. Known hypersensitivity or contraindication to cyclophosphamide
2. Known hypersensitivity or contraindications to Nivolumab or Ipilimumab.
3. Other malignancies, either simultaneous or within the last 2 years
4. Active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
5. Pregnancy and / or lactation
6. Patients who are sexually active refusing to use effective contraception (oral contraception, intrauterine devices, barrier method of contraception in conjunction with spermicidal jelly or surgical sterile)
7. Current or recent (within 4 weeks prior to start of trial treatment) treatment with another investigational drug or participation in another investigational trial
8. Severe concomitant diseases (e.g. immune deficiency syndrome)
9. Severe psychological disease or neurological damage without possibility to communicate
10. Clinical signs of intracranial pressure
11. Intracerebral hemorrhage, gliomatosis
12. No severe blood count abnormalities: leukocytes < 2.000/µl, Hb <10 g/dl, thrombocytes < 100.000/µl
13. No severe liver enzyme elevation (> 2-3x fold of normal)
14. Ongoing reirradiation or chemotherapy (within the last 4 weeks) (irradiation of formerly non-involved fields is allowed, but not part of this study)
15. Estimated life expectancy of less than 2 months
16. Preexisting severe cardiac disease
17. Presence of unresectable spinal metastases
18. Karnofsky index < 50%
19. Active infection within the last 2 weeks
20. Previous infection with Human Immunodeficiency, Hepatitis C, Human T-Lymphocyte 1/2, Hepatitis B Virus, Lues, protozoan parasites, or other chronic bacterial infections.
21. With regard to prevention of variant Creutzfeldt-Jakob disease the following patients have to be excluded.
22. Patients receiving systemic immunosuppressive or immunoactivating substances.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
6 month overall survival | 6 months
  overall survival 6 months after diagnosis of relapse

SECONDARY OUTCOMES:
overall survival | 12-24 months
  overall survival
progression-free survival | 12-24 months
  progression-free survival
toxicity metronomic cyclophosphamide | 12-24 months
  frequency of adverse events associated with metronomic cyclophosphamide
toxicitiy vaccine | 12-24 months
  frequency of adverse events associated with the vaccine
toxicity checkpoint blockade | 12-24 months
  frequency of AEs/SAEs associated with Nivolumab and/or Ipilimumab
Treg frequency | 12-24 months
  frequency of CD4+CD25+CD127- regulatory T cells under metronomic cyclophosphamide in % of CD3+
Treg numbers | 12-24 months
  absolute numbers of CD4+CD25+CD127- regulatory T cells under metronomic cyclophosphamide per µl blood
T-cell response | 12-24 months
  Interferon-gamma Cytotoxic T cell (CTL) assay
serum cytokine levels | 12-24 months
  Tru Culture cytokine array
correlation with histopathological tumor characteristics | 12-24 months
  correlation of outcome/immune response with histopathology etc.

CONTACTS AND LOCATIONS:
Overall Officials: Kramm Christof, MD, Study Chair — Children's Hospital, University Medical Center Göttingen
Locations (1):
- University Children's Hospital, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lohr M, Freitag B, Technau A, Krauss J, Monoranu CM, Rachor J, Lutz MB, Hagemann C, Kessler AF, Linsenmann T, Wolfl M, Ernestus RI, Engelhardt S, Gelbrich G, Schlegel PG, Eyrich M. High-grade glioma associated immunosuppression does not prevent immune responses induced by therapeutic vaccines in combination with Treg depletion. Cancer Immunol Immunother. 2018 Oct;67(10):1545-1558. doi: 10.1007/s00262-018-2214-0. Epub 2018 Jul 27. PMID 30054667
- [Result] Eyrich M, Schreiber SC, Rachor J, Krauss J, Pauwels F, Hain J, Wolfl M, Lutz MB, de Vleeschouwer S, Schlegel PG, Van Gool SW. Development and validation of a fully GMP-compliant production process of autologous, tumor-lysate-pulsed dendritic cells. Cytotherapy. 2014 Jul;16(7):946-64. doi: 10.1016/j.jcyt.2014.02.017. Epub 2014 May 13. PMID 24831836
- See also: homepage for patient and families — https://www.kinderkrebsinfo.de/fachinformationen/studienportal/